CLINICAL TRIAL: NCT01052571
Title: A Randomized, Prospective, Double-Blind, Equivalence, Controlled Evaluation of the Effectiveness of Transforaminal Epidural Injections in Lumbar Disc Herniation or Radiculitis With or Without Steroids
Brief Title: Evaluation of the Effectiveness of Transforaminal Epidural Injections in Lumbar Disc Herniation or Radiculitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pain Management Center of Paducah (Other)
Responsible Party: Principal Investigator, Laxmaiah Manchikanti, MD, Medical Director, Pain Management Center of Paducah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Protocol 24
Record Dates: First submitted 2010-01-18; First posted 2010-01-20 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Low Back Pain
Keywords: Chronic low back pain; Lumbar disc herniation; Lower extremity pain; Lumbar radiculitis; Local anesthetic; Steroid; Lumbar transforaminal epidural injection
MeSH Terms: conditions — Low Back Pain; Intervertebral Disc Displacement; Radiculopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Without Steroids (Active Comparator): Group I patients receiving lumbar transforaminal epidural injections with an injection of local anesthetic (lidocaine 1% or bupivacaine 0.25%
  Interventions: Procedure: lumbar transforaminal epidural injections
- steroids (Active Comparator): Group II patients will receive lumbar transforaminal epidural injections with 1% lidocaine or 0.25% bupivacaine with 3 mg of steroid per level
  Interventions: Procedure: lumbar transforaminal epidural injections

INTERVENTIONS:
Procedure: lumbar transforaminal epidural injections — with an injection of local anesthetic or with 1% lidocaine or 0.25% bupivacaine with 3 mg of steroid per level
  Other Names: Transforaminal Epidural

SUMMARY:
To evaluate differences in outcomes in patients receiving steroids compared to those patients randomized to the local anesthetic group who did not receive steroids.

To evaluate and compare the adverse event profile in all patients.

DETAILED DESCRIPTION:
Recruitment is indicated in patients with chronic low back and lower extremity pain secondary to lumbar disc herniation and/or lumbar radiculitis of at least 6-months duration, non-responsive to conservative management with NSAIDs, physical therapy, chiropractic treatment, and exercises.

This is a single center study performed in an interventional pain management referral center in the United States.

The study involves 120 patients studied in 2 groups with 60 patients in each group. Randomization includes sequence generation, allocation concealment, implementation, and blinding.

Data management analysis includes sample size justification of 40 patients in each group with a power of 80% and a 0.05% 2-sided significance level. Statistical methodology includes chi-squared statistics, Fisher's exact test, t-test, and paired t-test with significance evaluated at P value < 0.05.

ELIGIBILITY:
Inclusion criteria:

* Patients with disc herniation or radiculitis
* Patients who are 18 years of age
* Patients with a history of chronic function-limiting low back and lower extremity pain of at least 6 months duration
* Patients who are competent to understand the study protocol and provide voluntary, written informed consent and participate in outcome measurements

Exclusion criteria:

* Previous lumbar surgery, radiculitis secondary to spinal stenosis without disc herniation
* Uncontrollable or unstable opioid use
* Uncontrolled psychiatric disorders
* Uncontrolled medical illness either acute or chronic
* Any conditions that could interfere with the interpretation of the outcome assessments
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-02; Primary Completion 2012-01 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Numeric rating scale (NRS), Oswestry Disability Index (ODI), duration of significant pain relief, opioid intake, and return to work | Outcomes are measured at baseline and at 3, 6, 12, 18, and 24 months post-treatment.

SECONDARY OUTCOMES:
Adverse event profile of side effects and complications. | Adverse events are measured at baseline and at 3, 6, 12, 18, and 24 months post-treatment, and at any time during the procedure or after the procedure the adverse events are suspected or expected.

CONTACTS AND LOCATIONS:
Overall Officials: Laxmaiah Manchikanti, MD, Principal Investigator — Ambulatory Surgery Center, Paducah
Locations (1):
- Ambulatory Surgery Center, Paducah, Kentucky, United States